CLINICAL TRIAL: NCT01216358
Title: The Boston Migraine and Contraception Study
Brief Title: Boston Migraine and Contraception Study
Acronym: BMAC
Status: Completed | Type: Observational
Sponsor: Planned Parenthood League of Massachusetts (Other)
Collaborators: Brigham and Women's Hospital (Other); American Headache Society (Other); Society of Family Planning (Other)
Responsible Party: Sponsor
Other Study IDs: 2009P000464
Record Dates: First submitted 2010-10-06; First posted 2010-10-07 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: Headache
Keywords: Headache; Contraception
MeSH Terms: conditions — Headache

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Arm 1: Combined contraceptive: Initiating an estrogen/progesterone contraceptive
- Arm 2: Progesterone only contraceptive: Initiating a progesterone-only contraceptive
- Arm 3 (control): Non-hormonal contraceptive: Initiating or using non-hormonal contraception or not using contraception

SUMMARY:
The objectives of this prospective, descriptive study are to:

1. generate estimates of the incidence, prevalence, persistence, clinical impact and attributable risk of migraine due to hormonal contraception (HC) use; and
2. identify predictive factors for clinically significant changes in headache attributable to HC use.

The investigators hypothesize that:

1. Most women with pre-existing migraine will have no significant change from baseline headache frequency or clinical impact attributable to HC at 3 months following initiation; a minority will report clinically significant worsening or improvement
2. The incidence of headache and migraine in HC users will not be significantly different from their incidence in NHC users
3. There will be identifiable risk factors for development or worsening of headache/migraine in the minority of HC users where that occurs.

ELIGIBILITY:
Inclusion Criteria:

* Proficiency in English
* Medically eligible for her chosen form of contraception per standard PPLM clinic protocol
* (For Study Arm A) Desire initiation of an estrogen/progesterone contraceptive method at time of clinic presentation and evaluation
* (For Study Arm B) Desire initiation of a progesterone only contraceptive method at time of clinic presentation and evaluation
* (For Control Arm) Initiating a non-hormonal contraceptive, or not initiating any contraceptive method
* (For Control Arm) Stated intention of not initiating any hormonal contraception over the 3 month study period
* Agreeing to study procedures

Exclusion Criteria:

* Inability to speak and read English
* (For Control Arm) Use of hormonal contraceptive in the past 3 months
* (For Control Arm) Been pregnant in the past 3 months
* States an intention to discontinue use of their newly initiated contraceptive (or lack of contraceptive) before the end of the 3 month study period
* Unwilling or unable to comply with study follow-up procedures
* Inability to give informed consent
* Previous participation in this study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health female adults, patients of Planned Parenthood League of Massachusetts
Sampling Method: Non-Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2010-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Proportion of days with headache | 84 days
  Our primary outcome is the change in the proportion of headache days over 84 days, adjusted for baseline headache frequency

SECONDARY OUTCOMES:
Averages for percentage of headache days/28 days | 84 days
  Our secondary outcome will compare averages for the percentage of headache days/28 days for the days 1-28, days 29-56 and days 57-84, adjusted for baseline frequency

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, MD, Principal Investigator — Planned Parenthood League of Massachusetts
Locations (1):
- Planned Parenthood League of Massachusetts, Boston, Massachusetts, United States